CLINICAL TRIAL: NCT07231445
Title: A Phase Ib Study Evaluating the Safety and Efficacy of ZG006 in Combination With PD-1/PD-L1 Immune Checkpoint Inhibitors as First-Line Standard Therapy in Participants With Extensive Stage Small-Cell Lung Cancer
Brief Title: Study of ZG006 in Combination With PD-1/PD-L1 Immune Checkpoint Inhibitors as First-Line Standard Therapy in Participants With Extensive Stage Small-Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Suzhou Zelgen Biopharmaceuticals Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZG006-004
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part 1：Group A (Experimental): ZG006 D1: 1 mg; D22 onward: 10 mg; Q3W；Serplulimab 4.5 mg/kg，Q3W
  Interventions: Drug: ZG006; Drug: Serplulimab
- Part 1：Group B (Experimental): ZG006 D1: 1 mg; D22 onward: 30 mg; Q3W；Serplulimab 4.5 mg/kg，Q3W
  Interventions: Drug: ZG006; Drug: Serplulimab

INTERVENTIONS:
Drug: ZG006 — ZG006 will be administered as an IV infusion.
Drug: Serplulimab — Serplulimab will be administered as an IV infusion.

SUMMARY:
This is a randomized, multicenter, phase Ib study to evaluate the safety and efficacy of ZG006 combined with PD-1/PD-L1 immune checkpoint inhibitors (±chemotherapy) as first-line therapy in Participants with extensive stage small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants with histologically or cytologically confirmed ES-SCLC.
* Fully understand the study and voluntarily sign the informed consent form;
* Male or female 18~75 years of age;
* Eastern Cooperative Oncology Group(ECOG) Performance Status of 0 or 1;
* Life expectancy ≥ 3 months;

Exclusion Criteria:

* Participants were deemed unsuitable for participating in the study by the investigator for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-12-23 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Experiencing Dose-limiting toxicities (DLTs) | Up to Day 28
Number of Participants Experiencing Treatment-emergent Adverse Events (TEAEs) | Up to 2 Years

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 | Up to 2 Years
Maximum Serum Concentration (Cmax) of ZG006 | Up to 2 Years
Area Under the Concentration-time Curve (AUC) Over the Dosing Interval for ZG006 | Up to 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Jason Wu, Study Chair — Suzhou Zelgen Biopharmaceuticals Co.,Ltd
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China